CLINICAL TRIAL: NCT01164085
Title: Intravitreal Ketorolac for Chronic Uveitis:A Phase I Investigational Safety Study
Brief Title: Intravitreal Ketorolac for Chronic Uveitis: A Investigational Safety Study
Acronym: INCITE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Stephen J. Kim, MD, Principal Investigator, Vanderbilt University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 091196
Record Dates: First submitted 2010-04-19; First posted 2010-07-16 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Inflammation
Keywords: Inflammation; Macular Edema
MeSH Terms: conditions — Inflammation; Macular Edema | interventions — Tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketorolac (Experimental): 4mg intravitreal injection of ketorolac
  Interventions: Drug: Intravitreal Ketorolac

INTERVENTIONS:
Drug: Intravitreal Ketorolac — 4mg of intravitreal ketorolac
  Other Names: ketorolace, tromethamine, preservative free

SUMMARY:
Intraocular delivery of ketorolac will be an effective means to treat inflammation and macular edema and prevent structural complications and vision loss in patients with uveitis who are unable to tolerate corticosteroids due to their side effects.

DETAILED DESCRIPTION:
A Phase I safety study of intravitreal ketorolac in patients with chronic inflammation and complications due to inflammation who have either failed medical therapy or who cannot tolerate corticosteroids due to side effects.

Specific Aims

1. Test the safety of intraocular injection of 4mg of ketorolac in patients who have intractable uveitis or complications of uveitis such as chronic macular edema who are unable to tolerate corticosteroids due to their side effects.
2. Test the efficacy of intraocular 4m ketorolac of treating inflammation or structural complications of inflammation in patients with uveitis who are unable to tolerate corticosteroids due to their side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers
* Chronic intractable uveitis or chronic complications of uveitis (macular edema)despite maximal medical treatment
* Unable to tolerate corticosteroids due to side effects

Exclusion Criteria:

* 18 years or younger
* Have active ocular infection
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety | 90 days
  Baseline and 90 day electroretinogram and goldmann visual fields will be compared to assess for retinal toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Kim, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Eye Institute, Nashville, Tennessee, United States

REFERENCES:
- [Result] Kim SJ, Doherty TJ, Cherney EF. Intravitreal ketorolac for chronic uveitis and macular edema: a pilot study. Arch Ophthalmol. 2012 Apr;130(4):456-60. doi: 10.1001/archopthalmol.2011.2627. PMID 22491916
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/22491916